CLINICAL TRIAL: NCT04089787
Title: Shortened Antibiotic Treatment in Community-Acquired Pneumonia: A Nationwide Danish Randomized Controlled Trial
Brief Title: Shortened Antibiotic Treatment of 5 Days in Community-Acquired Pneumonia
Acronym: CAP5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Benfield (Other)
Responsible Party: Sponsor-Investigator, Thomas Benfield, Clinical Professor, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-19014479; 2019-000404-15 (EudraCT Number)
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-acquired pneumonia; Treatment duration; Pneumonia; Lung Diseases; Respiratory Tract Diseases; Respiratory Tract Infections; Bacterial Infections; Pneumonia, Bacterial; Anti-Infective Agents; Anti-Bacterial Agents
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia; Lung Diseases; Respiratory Tract Diseases; Respiratory Tract Infections; Bacterial Infections; Pneumonia, Bacterial | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Shortened antibiotic treatment of 5 days
  Interventions: Other: Intervention
- Control group (Active Comparator): Antibiotic treatment of 7 days or longer at the discretion of the treating physician
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — Shortened antibiotic treatment of 5 days
  Arms: Intervention group
Other: Control — Antibiotic treatment of 7 days or longer at the discretion of the treating physician
  Arms: Control group

SUMMARY:
CAP5 is an investigator-initiated multicentre non-inferiority randomized controlled trial which aims to assess the efficacy and safety of shortened antibiotic treatment duration of community-acquired pneumonia (CAP) in hospitalized adult patients based on clinical stability criteria.

Three to five days after initiation of antimicrobial therapy for CAP, participants are randomized 1:1 to parallel treatment arms: 5 days (intervention) or minimum 7 days (control) of antibiotic treatment. The intervention group discontinues antibiotics at day 5 if clinically stable and afebrile for at least 48 hours. The control group receives antibiotics for a duration of 7 days or longer at the discretion of the treating physician.

The primary outcome is 90-day survival which will be tested with a non-inferiority margin of 6%.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with community-acquired pneumonia; defined as new pulmonary infiltrate on chest X-ray and/or CT scan and at least one symptom compatible with pneumonia (cough, fever, dyspnoea and/or chest pain)
* Initiation of antibiotics within 12 hours of the time of the chest X-ray with an infiltrate
* Age ≥ 18 years
* Afebrile (temperature ≤ 37.8 °C) for 48 hours at randomization
* Clinically stable at randomization (systolic blood pressure ≥ 90 mm Hg, heart rate ≤ 100/min., respiratory rate ≤ 24/min., peripheral oxygen saturation ≥ 90%)

Exclusion Criteria:

* Immunosuppression (HIV-positive, neutropenia, corticosteroid treatment (≥10 mg/day of prednisone or the equivalent for >30 days), chemotherapy, immunosuppressive agents, immunosuppressed after solid organ transplantation, asplenia)
* Hospitalization during the previous 14 days
* Antibiotic treatment (>2 days) within the past 30 days, directed at lower respiratory tract pathogens
* Uncommon cause requiring longer duration of antimicrobial therapy (Pseudomonas aeruginosa, Staphylococcus aureus, Mycobacterium spp., fungi)
* Extrapulmonary infection (e.g. endocarditis, meningitis, or abscess)
* Pleural empyema or lung abscess
* Pleural effusion requiring drainage tube
* Intensive care unit (ICU) admittance
* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
90-day survival | within 90 days

SECONDARY OUTCOMES:
Duration of antibiotic treatment | within 90 days
  Days that the participant receives antibiotic treatment for pneumonia, adding intravenous and oral therapy
Length of hospital stay | within 90 days
  Days from the date of hospital admission for pneumonia to the date of discharge
Antibiotic adverse events | within 90 days
  Number of participants with adverse events with possible relation to the antibiotic treatment of pneumonia
Serious adverse events | within 90 days
  Number of participants with serious adverse events according to International Council of Harmonisation-Good Clinical Practice (ICH-GCP) guidelines
Major complications | within 90 days
  Number of participants with major complications, including pleural effusion, pleural empyema, lung abscess, respiratory failure, severe sepsis, renal failure, use of non-invasive or invasive ventilation, need for vasopressors, and intensive care unit (ICU) admission
Use of antimicrobials after discharge | within 90 days
  Days of antibiotic treatment for any reason after hospital discharge
Post-discharge follow-up visits | within 90 days
  Number of participants with medical visits after hospital discharge, including visits at the outpatient clinic and at the general practitioner
Readmissions | days 30 and 90
  Number of participants with readmissions for reasons related to or unrelated to pneumonia
Mortality | in-hospital, days 30 and 90
  Number of deaths by any cause

CONTACTS AND LOCATIONS:
Overall Officials: Simone Bastrup Israelsen, MD, Principal Investigator — Copenhagen University Hospital - Amager and Hvidovre, Hvidovre, Denmark
Locations (7):
- Denmark (7):
  - Aalborg University Hospital, Aalborg
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Hospital, Gentofte Municipality
  - Herlev Hospital, Herlev
  - Nordsjællands Hospital, Hillerød
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No
Trial data will be made available in anonymous form at public clinical trial databases when the trial has ended. Anonymized patient-level data and other detailed information will be provided by reasonable request to the principal investigator.

REFERENCES:
- [Background] Welte T, Torres A, Nathwani D. Clinical and economic burden of community-acquired pneumonia among adults in Europe. Thorax. 2012 Jan;67(1):71-9. doi: 10.1136/thx.2009.129502. Epub 2010 Aug 20. PMID 20729232
- [Background] Ramirez JA, Wiemken TL, Peyrani P, Arnold FW, Kelley R, Mattingly WA, Nakamatsu R, Pena S, Guinn BE, Furmanek SP, Persaud AK, Raghuram A, Fernandez F, Beavin L, Bosson R, Fernandez-Botran R, Cavallazzi R, Bordon J, Valdivieso C, Schulte J, Carrico RM; University of Louisville Pneumonia Study Group. Adults Hospitalized With Pneumonia in the United States: Incidence, Epidemiology, and Mortality. Clin Infect Dis. 2017 Nov 13;65(11):1806-1812. doi: 10.1093/cid/cix647. PMID 29020164
- [Background] Egelund GB, Jensen AV, Andersen SB, Petersen PT, Lindhardt BO, von Plessen C, Rohde G, Ravn P. Penicillin treatment for patients with Community-Acquired Pneumonia in Denmark: a retrospective cohort study. BMC Pulm Med. 2017 Apr 20;17(1):66. doi: 10.1186/s12890-017-0404-8. PMID 28427381
- [Background] Uranga A, Espana PP, Bilbao A, Quintana JM, Arriaga I, Intxausti M, Lobo JL, Tomas L, Camino J, Nunez J, Capelastegui A. Duration of Antibiotic Treatment in Community-Acquired Pneumonia: A Multicenter Randomized Clinical Trial. JAMA Intern Med. 2016 Sep 1;176(9):1257-65. doi: 10.1001/jamainternmed.2016.3633. PMID 27455166
- [Background] Aliberti S, Ramirez J, Giuliani F, Wiemken T, Sotgiu G, Tedeschi S, Carugati M, Valenti V, Marchioni M, Camera M, Piro R, Del Forno M, Milani G, Faverio P, Richeldi L, Deotto M, Villani M, Voza A, Tobaldini E, Bernardi M, Bellone A, Bassetti M, Blasi F. Individualizing duration of antibiotic therapy in community-acquired pneumonia. Pulm Pharmacol Ther. 2017 Aug;45:191-201. doi: 10.1016/j.pupt.2017.06.008. Epub 2017 Jun 27. PMID 28666965
- [Background] Dunbar LM, Wunderink RG, Habib MP, Smith LG, Tennenberg AM, Khashab MM, Wiesinger BA, Xiang JX, Zadeikis N, Kahn JB. High-dose, short-course levofloxacin for community-acquired pneumonia: a new treatment paradigm. Clin Infect Dis. 2003 Sep 15;37(6):752-60. doi: 10.1086/377539. Epub 2003 Aug 28. PMID 12955634
- [Background] el Moussaoui R, de Borgie CA, van den Broek P, Hustinx WN, Bresser P, van den Berk GE, Poley JW, van den Berg B, Krouwels FH, Bonten MJ, Weenink C, Bossuyt PM, Speelman P, Opmeer BC, Prins JM. Effectiveness of discontinuing antibiotic treatment after three days versus eight days in mild to moderate-severe community acquired pneumonia: randomised, double blind study. BMJ. 2006 Jun 10;332(7554):1355. doi: 10.1136/bmj.332.7554.1355. PMID 16763247
- [Background] Torres A, Muir JF, Corris P, Kubin R, Duprat-Lomon I, Sagnier PP, Hoffken G. Effectiveness of oral moxifloxacin in standard first-line therapy in community-acquired pneumonia. Eur Respir J. 2003 Jan;21(1):135-43. doi: 10.1183/09031936.03.00045202. PMID 12570122
- [Background] File TM Jr, Mandell LA, Tillotson G, Kostov K, Georgiev O. Gemifloxacin once daily for 5 days versus 7 days for the treatment of community-acquired pneumonia: a randomized, multicentre, double-blind study. J Antimicrob Chemother. 2007 Jul;60(1):112-20. doi: 10.1093/jac/dkm119. Epub 2007 May 30. PMID 17537866
- [Background] Tamma PD, Avdic E, Li DX, Dzintars K, Cosgrove SE. Association of Adverse Events With Antibiotic Use in Hospitalized Patients. JAMA Intern Med. 2017 Sep 1;177(9):1308-1315. doi: 10.1001/jamainternmed.2017.1938. PMID 28604925
- [Background] Huttner A, Harbarth S, Carlet J, Cosgrove S, Goossens H, Holmes A, Jarlier V, Voss A, Pittet D. Antimicrobial resistance: a global view from the 2013 World Healthcare-Associated Infections Forum. Antimicrob Resist Infect Control. 2013 Nov 18;2:31. doi: 10.1186/2047-2994-2-31. eCollection 2013. PMID 24237856
- [Background] Pollack LA, Srinivasan A. Core elements of hospital antibiotic stewardship programs from the Centers for Disease Control and Prevention. Clin Infect Dis. 2014 Oct 15;59 Suppl 3(Suppl 3):S97-100. doi: 10.1093/cid/ciu542. PMID 25261548
- [Background] Madaras-Kelly KJ, Burk M, Caplinger C, Bohan JG, Neuhauser MM, Goetz MB, Zhang R, Cunningham FE; Pneumonia Duration of Therapy Medication Utilization Evaluation Group. Total duration of antimicrobial therapy in veterans hospitalized with uncomplicated pneumonia: Results of a national medication utilization evaluation. J Hosp Med. 2016 Dec;11(12):832-839. doi: 10.1002/jhm.2648. Epub 2016 Aug 16. PMID 27527659
- [Background] Aliberti S, Blasi F, Zanaboni AM, Peyrani P, Tarsia P, Gaito S, Ramirez JA. Duration of antibiotic therapy in hospitalised patients with community-acquired pneumonia. Eur Respir J. 2010 Jul;36(1):128-34. doi: 10.1183/09031936.00130909. Epub 2009 Nov 19. PMID 19926738
- [Background] Li JZ, Winston LG, Moore DH, Bent S. Efficacy of short-course antibiotic regimens for community-acquired pneumonia: a meta-analysis. Am J Med. 2007 Sep;120(9):783-90. doi: 10.1016/j.amjmed.2007.04.023. PMID 17765048
- [Background] Dimopoulos G, Matthaiou DK, Karageorgopoulos DE, Grammatikos AP, Athanassa Z, Falagas ME. Short- versus long-course antibacterial therapy for community-acquired pneumonia : a meta-analysis. Drugs. 2008;68(13):1841-54. doi: 10.2165/00003495-200868130-00004. PMID 18729535
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Background] Schrag SJ, Pena C, Fernandez J, Sanchez J, Gomez V, Perez E, Feris JM, Besser RE. Effect of short-course, high-dose amoxicillin therapy on resistant pneumococcal carriage: a randomized trial. JAMA. 2001 Jul 4;286(1):49-56. doi: 10.1001/jama.286.1.49. PMID 11434826
- [Background] Chastre J, Wolff M, Fagon JY, Chevret S, Thomas F, Wermert D, Clementi E, Gonzalez J, Jusserand D, Asfar P, Perrin D, Fieux F, Aubas S; PneumA Trial Group. Comparison of 8 vs 15 days of antibiotic therapy for ventilator-associated pneumonia in adults: a randomized trial. JAMA. 2003 Nov 19;290(19):2588-98. doi: 10.1001/jama.290.19.2588. PMID 14625336
- [Background] File TM Jr. Clinical efficacy of newer agents in short-duration therapy for community-acquired pneumonia. Clin Infect Dis. 2004 Sep 1;39 Suppl 3:S159-64. doi: 10.1086/421354. PMID 15546111
- [Background] Guillemot D, Carbon C, Balkau B, Geslin P, Lecoeur H, Vauzelle-Kervroedan F, Bouvenot G, Eschwege E. Low dosage and long treatment duration of beta-lactam: risk factors for carriage of penicillin-resistant Streptococcus pneumoniae. JAMA. 1998 Feb 4;279(5):365-70. doi: 10.1001/jama.279.5.365. PMID 9459469
- [Background] Halm EA, Fine MJ, Marrie TJ, Coley CM, Kapoor WN, Obrosky DS, Singer DE. Time to clinical stability in patients hospitalized with community-acquired pneumonia: implications for practice guidelines. JAMA. 1998 May 13;279(18):1452-7. doi: 10.1001/jama.279.18.1452. PMID 9600479
- [Background] Menendez R, Torres A, Rodriguez de Castro F, Zalacain R, Aspa J, Martin Villasclaras JJ, Borderias L, Benitez Moya JM, Ruiz-Manzano J, Blanquer J, Perez D, Puzo C, Sanchez-Gascon F, Gallardo J, Alvarez CJ, Molinos L; Neumofail Group. Reaching stability in community-acquired pneumonia: the effects of the severity of disease, treatment, and the characteristics of patients. Clin Infect Dis. 2004 Dec 15;39(12):1783-90. doi: 10.1086/426028. Epub 2004 Nov 18. PMID 15578400
- [Background] Choudhury G, Mandal P, Singanayagam A, Akram AR, Chalmers JD, Hill AT. Seven-day antibiotic courses have similar efficacy to prolonged courses in severe community-acquired pneumonia--a propensity-adjusted analysis. Clin Microbiol Infect. 2011 Dec;17(12):1852-8. doi: 10.1111/j.1469-0691.2011.03542.x. Epub 2011 Sep 15. PMID 21919994
- [Derived] Israelsen SB, Tingsgard S, Thorlacius-Ussing L, Knudsen A, Lindegaard B, Johansen IS, Mygind LH, Ravn P, Benfield T. Short-course antibiotic therapy of 5 days in community-acquired pneumonia (CAP5): study protocol for a randomised controlled trial. BMJ Open. 2023 Jul 21;13(7):e069013. doi: 10.1136/bmjopen-2022-069013. PMID 37479519

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT04089787/SAP_000.pdf